CLINICAL TRIAL: NCT03657342
Title: A Phase III Clinical Trial to Demonstrate Efficacy / Safety of Liposomal Cyclosporine A + Standard of Care (SoC) vs SoC Alone in Treating Chronic Lung Allograft Dysfunction / Bronchiolitis Obliterans in Patients Post Single Lung Transplant
Brief Title: Efficacy + Safety of Liposome Cyclosporine A to Treat Bronchiolitis Obliterans Post Single Lung Transplant (BOSTON-1)
Acronym: BOSTON-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zambon SpA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BT - L-CsA - 301 - SLT; 2018-003204-39 (EudraCT Number)
Record Dates: First submitted 2018-08-30; First posted 2018-09-05 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Bronchiolitis Obliterans; Chronic Rejection of Lung Transplant; Lung Transplant Rejection; Lung Transplant; Complications; Lung Transplant Failure and Rejection; Chronic Lung Allograft Dysfunction
MeSH Terms: conditions — Bronchiolitis Obliterans; Rejection, Psychology | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: This was an open-label clinical trial. Clinical trial monitors, treating physicians, study nurses, study coordinators, and enrolled patients were not blinded to treatment assignment.
  However, the pulmonary function technicians, respiratory therapists, or physiotherapists who conducted spirometry on-site were blinded to treatment assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-CsA treatment plus SoC (Experimental): Liposomal Cyclosporine A 5 mg twice daily for 48 weeks + Standard of Care Therapy
  Interventions: Drug: Liposomal Cyclosporine A
- Control treatment (Active Comparator): In this arm only the standard of care is administered. Standard of care is a maintenance regimen of immunosuppressive agents.
  Interventions: Drug: standard of care

INTERVENTIONS:
Drug: Liposomal Cyclosporine A — This formulation is developed for inhalation use and delivered via the PARI eFlow® Device, which is a new technology of nebulizing liquid drugs with a perforated vibrating membrane resulting in an aerosol with a low ballistic momentum and a high percentage of droplets in a respirable size range of 3-5 μm
  Other Names: L-CsA
  Arms: L-CsA treatment plus SoC
Drug: standard of care — Standard of Care Therapy. Eligible patients should be on a maintenance regimen of immunosuppressive agents including tacrolimus, a second agent such as but not limited to MMF or azathioprine, and a systemic corticosteroid such as prednisone as third agent. The regimen must be stable within 4 weeks prior to randomization with respect to the therapeutic agents. Patients receiving azithromycin for prophylaxis or treatment of BOS, must be on a stable regimen for a least 4-weeks prior to randomization and will continue to receive azithromycin during the trial as deemed appropriate by the investigator.
  Other Names: SoC
  Arms: Control treatment

SUMMARY:
The objective of this trial is to assess the efficacy and safety of aerosolized liposomal cyclosporine A (L-CsA) as add-on therapy to standard of care (SoC) as compared to SoC alone in single lung transplant recipients with chronic lung allograft dysfunction (CLAD)-bronchiolitis obliterans syndrome (BOS).

DETAILED DESCRIPTION:
BOSTON-1 was a Phase III, prospective, multicenter, randomized, open-label, controlled clinical trial of L-CsA for the treatment of BOS in adults diagnosed with CLAD-BOS following single lung transplant.

Eligible patients were randomized to receive either L-CsA (5 mg) via the PARI eFlow® Device (L-CsA eFlow) twice daily plus SoC treatment or SoC alone for a period of 48 weeks.

Regardless of treatment allocation, all patients continued to receive their SoC regimen for maintenance of the lung allograft. Maintenance immunosuppressive therapy including tacrolimus, a second agent such as, but not limited to, MMF or azathioprine, and a systemic corticosteroid such as prednisone as third agent was administered according to institutional standards.

Up to 11 study visits (screening, V1 through V10) were planned. Spirometry was measured at all visits according to American Thoracic Society/European Respiratory Society 2005 guidelines. Spirometry measurements on-site were performed by pulmonary function technicians, respiratory therapists, or physiotherapists who were blinded to each patient's study treatment assignment.

Safety assessments at every study visit included physical examination, vital signs, adverse event (AE) reporting, and clinical laboratory tests. Acute tolerability of L-CsA was assessed by spirometry before and 1 hour and 4 hours after inhalation of L-CsA at initial dosing.

All patients who completed the study were eligible to continue in an open-label extension trial of L-CsA (BOSTON-3 [Study BT-L-CsA-303-FU]).

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients ≥ 18 years who received a single lung transplant at least 12 months prior to Screening.
2. Patients with BOS diagnosis defined as CLAD-BOS phenotype with:

   1. Screening FEV1 between 85-51% of personal best FEV1 value post-transplant OR
   2. Screening FEV1 >85% of personal best FEV1 associated with EITHER a ≥ 200 mL decrease in FEV1 in the previous 12 months OR according to medical history showing BOS progression.
3. Diagnosis of CLAD-BOS must have been made at least 12 months after lung transplantation and

   1. within 12 months prior to the screening visit OR
   2. more than 12 months from screening and patient must have shown a decline in FEV1 ≥ 200ml in the previous 12 months before screening, which was not due to acute infection or acute organ rejection.
4. Patients in whom the diagnosis of BOS had been confirmed by the elimination of other possible causes of obstructive or restrictive lung disease (CLAD - RAS phenotype, see Protocol Specific Definitions).
5. Patients should have been on a maintenance regimen of immunosuppressive agents including tacrolimus, a second agent such as but not limited to mycophenolate mofetil (MMF) or azathioprine, and a systemic corticosteroid such as prednisone as third agent. The regimen must have been stable within 4 weeks prior to randomization with respect to the therapeutic agents. In case a patient was also receiving concomitant azithromycin for prophylaxis or treatment of BOS in addition to the previously described immunosuppressive regimen, azithromycin must have been on a stable regimen for at least 4 weeks prior to randomization.
6. Patients capable of understanding the purposes and risks of the clinical trial, who had given written informed consent and agreed to comply with the clinical trial requirements/visit schedules, and who were capable of aerosol inhalation. Patients must have consented to retrieve prespecified data from the historic medical record (e.g., information related to the transplant surgery; spirometry data; medication use).
7. Women of childbearing potential must have had a negative serum or urine pregnancy test within 7 days prior to randomization and must agree to use one of the methods of contraception listed in Appendix II of the Protocol through their End of Study (EoS) Visit.
8. Patients had no concomitant diagnoses that were considered fatal within one year (12 months) of Screening.

Exclusion Criteria:

1. Patients with confirmed other causes for loss of lung function, such as acute infection, acute rejection, restrictive allograft syndrome (CLAD - RAS phenotype, see Protocol Specific Definition ), etc.
2. Patients with acute antibody-mediated rejection at Screening. In this context, clinically stable patients (as judged by the Investigator) with detectable levels of donor specific antibodies (DSA) at the Screening Visit were eligible for the study.
3. Active acute bacterial, viral, or fungal infection not successfully resolved at least 4 weeks prior to the Screening Visit. Patients with chronic infection or colonization who were clinically stable as per judgement of the Investigator are eligible for the study.
4. Mechanical ventilation (including CPAP) within 12 weeks prior to Randomization.
5. Patients with uncontrolled hypertension.
6. Patient had baseline resting oxygen saturation of < 89% on room air or use of supplemental oxygen at rest.
7. Evidence of functional airway stenosis (e.g., bronchomalacia/tracheomalacia, airway stents, or airways requiring balloon dilatations to maintain patency) with onset after the initial diagnosis of BOS and ongoing at Screening and/or Baseline Visit.
8. Known hypersensitivity to L-CsA or to cyclosporine A.
9. Patients with chronic renal failure, defined as serum creatinine > 2.5 mg/dL at screening, or requiring chronic dialysis.
10. Patients with liver disease and serum bilirubin > 3-fold upper limit of normal range or transaminases > 2.5 upper limit of normal range.
11. Patients with active malignancy within the previous 2 years, including post-transplant lymphoproliferative disorder, with the exception of treated, localized basal and squamous cell carcinomas.
12. Pregnant women or women who were unwilling to use appropriate birth control to avoid pregnancy through their End of Study (EoS) Visit.
13. Women who were currently breastfeeding.
14. Receipt of an investigational drug as part of a clinical trial within 4 weeks prior to the Screening Visit. This was defined as any treatment that was implemented under an Investigational New Drug (IND) or compassionate use.
15. Patients who had received extracorporeal photophoresis (ECP) for treatment of BOS within 1 month prior to Randomization.
16. Patients who were currently participating in an interventional clinical trial.
17. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary procedures.
18. Any co-existing medical condition that in the Investigator's judgment would substantially increase the risk associated with the patient's participation in the clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-03-26 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paola Castellani, MD, Study Director — Zambon SpA, Chief Medical Officer and R&D
Locations (39):
- United States (25):
  - Banner Health, Phoenix, Arizona
  - Norton Thoracic Institute at St. Joseph's Hospital, Phoenix, Arizona
  - UCLA Medical Center, Los Angeles, California
  - Stanford University Hospital, Palo Alto, California
  - UC San Francisco, San Francisco, California
  - University of Florida Medical Center, Gainesville, Florida
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Indiana University Health Methodist Hospital, Indianapolis, Indiana
  - University of Kentucky Albert B. Chandler Hospital, Lexington, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University Hospital, Baltimore, Maryland
  - 110, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - 113, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - 119, Columbus, Ohio
  - 108, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor University Medical Center, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor St. Luke's Medical Center, Houston, Texas
  - Houston Methodist Hospital, Houston, Texas
- Universitair Ziekenhuis Leuven, Leuven, Belgium
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France
- Germany (2):
  - Hannover Medical School - MHH Klinik für Pneumologie, Hanover
  - LMU Klinikum Großhadern, Munich
- Rabin Medical Center, Petah Tikva, Israel
- Spain (7):
  - Complexo Hospitalario de A Coruna, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Marques de Valdecilla, Santander
  - Hospital Universitario y Politécnico La Fe, Valencia
- United Kingdom (2):
  - Royal Papworth Hospital NHS Foundation Trust, Cambridge
  - University Hospital of South Manchester NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study randomized 62 patients globally from 26Mar2019 to 16Apr2024.
Pre-assignment Details: Of the 97 patients screened (up to 4 weeks screening period prior to Visit 1), 62 patients were enrolled, randomized, and treated.
Groups:
- SoC alone: In this control arm only the standard of care is administered. Standard of care is a maintenance regimen of immunosuppressive agents.
  standard of care: Standard of Care Therapy. Eligible patients should be on a maintenance regimen of immunosuppressive agents including tacrolimus, a second agent such as but not limited to MMF or azathioprine, and a systemic corticosteroid such as prednisone as third agent. The regimen must be stable within 4 weeks prior to randomization with respect to the therapeutic agents. Patients receiving azithromycin for prophylaxis or treatment of BOS, must be on a stable regimen for a least 4-weeks prior to randomization and will continue to receive azithromycin during the trial as deemed appropriate by the investigator.
Period: Overall Study
Arm/Group | L-CsA treatment plus SoC | SoC alone
Started | 32 | 30
FAS | 32 | 30
SAF | 32 | 30
PPS | 21 | 19
Completed | 20 | 23
Not Completed | 12 | 7
Not completed — Adverse Event, including SAE/Death | 6 | 3
Not completed — Withdrawal by Subject | 4 | 4
Not completed — PATIENT WITHDRAWN BY THE SPONSOR DUE TO USE OF CYCLOSPORINE A DURING TRIAL (NOT ALLOWED) | 1 | 0
Not completed — PI WITHDREW PATIENT DUE TO THE HIS/HER UNSTABLE CLINICAL CONDITION | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- L-CsA treatment plus SoC (SAF): Liposomal Cyclosporine A 5 mg twice daily for 48 weeks + Standard of Care Therapy
  Liposomal Cyclosporine A: This formulation is developed for inhalation use and delivered via the PARI eFlow® Device, which is a new technology of nebulizing liquid drugs with a perforated vibrating membrane resulting in an aerosol with a low ballistic momentum and a high percentage of droplets in a respirable size range of 3-5 μm
- SoC alone (SAF): In this control arm only the standard of care is administered. Standard of care is a maintenance regimen of immunosuppressive agents.
  standard of care: Standard of Care Therapy. Eligible patients should be on a maintenance regimen of immunosuppressive agents including tacrolimus, a second agent such as but not limited to MMF or azathioprine, and a systemic corticosteroid such as prednisone as third agent. The regimen must be stable within 4 weeks prior to randomization with respect to the therapeutic agents. Patients receiving azithromycin for prophylaxis or treatment of BOS, must be on a stable regimen for a least 4-weeks prior to randomization and will continue to receive azithromycin during the trial as deemed appropriate by the investigator.
- Total: Total of all reporting groups
Arm/Group | L-CsA treatment plus SoC (SAF) | SoC alone (SAF) | Total
Number analyzed (Participants) | 32 | 30 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 5 | 14
  >=65 years | 23 | 25 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (7.20) | 69.3 (5.28) | 68.0 (6.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 22 | 17 | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 29 | 29 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 28 | 25 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 21 | 20 | 41
  United Kingdom | 1 | 2 | 3
  Israel | 2 | 4 | 6
  Germany | 3 | 0 | 3
  Spain | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in FEV1 (L) From Baseline to Week 48
Description: FEV1 is the Forced Expiratory Volume in One Second. For FEV1 were considered primary the data collected from the on site COMPACT study spirometer. Baseline is the mean of the best FEV1 obtained with the study spirometer at Screening Visit and the pre-randomization best FEV1 obtained at the Baseline Visit (V1).The primary efficacy analysis was carried out using a Linear Mixed Model (LMM) for repeated measures, using all observed available FEV1 measurements. In case of death or re-transplantation events, FEV1 was imputed as zero at each nominal day post event.
  PS: Estimates are from a LMM on the response variable with factors for time splines, treatment, the interactions of time splines by treatment, baseline FEV1, the interactions of time splines with baseline FEV1, region, underlying indication for lung transplant (COPD vs all others), use of azithromycin at randomization, and time as random effect.
Time Frame: Week 48 (V9)
Population: FAS: The FAS is defined as all randomized patients. Patients were analyzed according to the treatment group to which they were randomized. All primary and secondary endpoints were performed using the FAS, unless otherwise specified. n=25 is the number of patients with data available, not the number of patients in the analysis set (N).
Measure: Least Squares Mean (Standard Error); unit: liters
Groups:
- L-CsA treatment plus SoC (FAS): Liposomal Cyclosporine A 5 mg twice daily for 48 weeks + Standard of Care Therapy
  Liposomal Cyclosporine A: This formulation is developed for inhalation use and delivered via the PARI eFlow® Device, which is a new technology of nebulizing liquid drugs with a perforated vibrating membrane resulting in an aerosol with a low ballistic momentum and a high percentage of droplets in a respirable size range of 3-5 μm
- SoC alone (FAS): In this control arm only the standard of care is administered. Standard of care is a maintenance regimen of immunosuppressive agents.
  standard of care: Standard of Care Therapy. Eligible patients should be on a maintenance regimen of immunosuppressive agents including tacrolimus, a second agent such as but not limited to MMF or azathioprine, and a systemic corticosteroid such as prednisone as third agent. The regimen must be stable within 4 weeks prior to randomization with respect to the therapeutic agents. Patients receiving azithromycin for prophylaxis or treatment of BOS, must be on a stable regimen for a least 4-weeks prior to randomization and will continue to receive azithromycin during the trial as deemed appropriate by the investigator.
Arm/Group | L-CsA treatment plus SoC (FAS) | SoC alone (FAS)
Number analyzed (Participants) | 25 | 25
liters | -0.186 (0.3093) | -0.090 (0.2879)
Statistical Analysis 1: Comparison: L-CsA treatment plus SoC (FAS) vs SoC alone (FAS); at V9; Test type: Superiority; p = 0.7310, Mixed Models Analysis — 1-sided p value; LS Mean Difference = -0.095, 95% CI 2-sided [-0.405 to 0.214]

2. Secondary Outcome: Mean Change in FEV1/FVC From Baseline to Week 48
Description: Forced Expiratory Volume in One Second on Forced Vital Capacity. It was analysed in the FAS using a LMM for repeated measurements and COMPACT data, with baseline FEV1/FVC among covariates. In case of death or re- transplantation events, FEV1/FVC was imputed as zero at each nominal day post event. FEV1/FVC is a calculated ratio used to diagnose obstructive and restrictive lung disease. It represents the proportion of a patient's vital capacity that he/she is able to expire in the first second of forced expiration to the full forced vital capacity.
Time Frame: Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ratio
Arm/Group | L-CsA treatment plus SoC (SAF) | SoC alone (SAF)
Number analyzed (Participants) | 25 | 25
ratio | 0.093 (0.2353) | 0.157 (0.2433)
Statistical Analysis 1: Comparison: L-CsA treatment plus SoC (SAF) vs SoC alone (SAF); Estimates were from a Linear Mixed Model on the response variable change from baseline in FEV1/FVC with factors for time splines, treatment, the interactions of time splines by treatment, baseline FEV1/FVC, the interactions of time splines with baseline FEV1/FVC, region (North America versus all other countries together), underlying indication for lung transplant (COPD versus all others), use of azithromycin at randomization, and time as random effect; Test type: Superiority; p = 0.8041, Mixed Models Analysis — 1-sided p value; least suare mean difference = -0.064, 95% CI 2-sided [-0.212 to 0.084]

3. Secondary Outcome: Time to Progression of Bronchiolitis Obliterans Syndrome (BOS)
Description: The progression of BOS is defined as the earliest of the following:
  * Absolute decrease from baseline in FEV1 by at least 10% or 200 mL and a decrease in FEV1/FVC by at least 5% (if a patient had an event that met this criterion for progression of BOS, progression of BOS must have been confirmed by measurements that were taken with COMPACT spirometer at least 2 weeks apart) OR
  * Worsening of BOS grade, OR
  * Re-transplantation, OR
  * Death from respiratory failure. Rules for censoring progression of BOS are set. More than one type of event might correspond to the event of BOS progression (even those occurring on the same date). In case progression of BOS was defined by more than one criterion on different dates, the earliest event date was considered, i.e., the date closer to randomization was used as the progression date.
Time Frame: From date of randomization until the date of first documented progression of BOS, or date of retransplantation, or date of death from respiratory failure, whichever came first, assessed up to 48 weeks.
Population: FAS: The FAS is defined as all randomized patients. Patients were analyzed according to the treatment group to which they were randomized. All primary and secondary endpoints were performed using the FAS, unless otherwise specified.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | L-CsA treatment plus SoC (FAS) | SoC alone (FAS)
Number analyzed (Participants) | 32 | 30
Weeks | NA [NA to NA] — Median and confidence interval limits were not achieved due to low number of events. | NA [NA to NA] — Median and confidence interval limits were not achieved due to low number of events.
Statistical Analysis 1: Comparison: L-CsA treatment plus SoC (FAS) vs SoC alone (FAS); Test type: Superiority; p = 0.1559, Regression, Cox — 1-sided p value. Adjusted Hazard Ratio calculated using Cox proportional hazards model with covariates of Treatment, Baseline FEV1, with Efron's method of tie handling; adjusted hazard ratio = 2.601, 95% CI 2-sided [0.408 to 16.585]

4. Other Pre Specified Outcome: Number of Patients With Adverse Events (AE)
Description: An AE is an untoward medical occurrence after exposure to a medicine, which is not necessarily caused by that medicine.
Time Frame: Baseline through study completion (week 48)
Population: SAF: The SAF was defined as all randomized patients receiving SoC and/or at least one dose of L-CsA, independently of the treatment allocation at randomization. All safety and tolerability data were summarized and analyzed using the SAF.
Measure: Count of Participants; unit: Participants
Arm/Group | L-CsA treatment plus SoC (SAF) | SoC alone (SAF)
Number analyzed (Participants) | 32 | 30
Participants
  No of patients with any AE | 32 | 25
  No. of patients with any TEAE leading to discontinuation of study treatment | 8 | 2
  No. of patients with any TEAE leading to study discontinuation | 6 | 3
  No. of patients with any TEAE leading to death | 6 | 3
  No. of patients with any TEAE of Grade 1 severity (Mild) | 22 | 22
  No. of patients with any TEAE of Grade 2 severity (Moderate) | 14 | 12
  No. of patients with any TEAE of Grade 3 severity (severe) | 15 | 8
  No. of patients with any study treatment-related TEAE | 11 | NA
  No. of patients with any serious TEAE | 20 | 14
  No. of patients with any serious treatment-related TEAE | 3 | NA

5. Other Pre Specified Outcome: Acute Tolerability of L-CsA: Change From Pre-dose to 1 hr and 4h Post-dose
Description: Acute tolerability of IMP (L-CsA) during initial dosing was determined by measuring spirometry 1 hour and 4 hours after treatment. The FEV1 was measured prior to dosing with L-CsA. A decline of ≥20% associated with symptoms could have warranted IMP discontinuation. Parameters reflecting acute tolerability of IMP were: spirometry, cough, or dyspnea.
Time Frame: Baseline through study completion Week 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | L-CsA treatment plus SoC (SAF)
Number analyzed (Participants) | 29
Liters
  1 hr Post-dose | -0.022 (0.0663)
  4 hr Post-dose | -0.019 (0.0701)

ADVERSE EVENTS:
Time Frame: Permanent assessment throughout the complete clinical trial period, from baseline (Week 0, Day 1, V1) till week 48 (V9)
Arm/Group | L-CsA treatment plus SoC (SAF) | SoC alone (SAF)
All-Cause Mortality (participants affected / at risk) | 6/32 | 3/30
Serious Adverse Events (participants affected / at risk) | 20/32 | 14/30
Other Adverse Events (participants affected / at risk) | 28/32 | 17/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-CsA treatment plus SoC (SAF) (N=32) | SoC alone (SAF) (N=30)
COVID-19 (Infections and infestations) | 7 (9) | 5 (5)
COVID-19 pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pneumonia pseudomonal (Infections and infestations) | 2 (3) | 0 (0)
Septic shock (Infections and infestations) | 2 (2) | 0 (0)
Clostridial sepsis (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0)
Parainfluenzae virus infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia pneumococcal (Infections and infestations) | 1 (1) | 0 (0)
Pseudomonal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Streptococcal sepsis (Infections and infestations) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 1 (1) | 0 (0)
Cytomegalovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (3) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 1 (1) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular failure (Cardiac disorders) | 0 (0) | 1 (1)
Multiple organ dysfunction syndrome (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 3 (4) | 0 (0)
Lung transplant rejection (Immune system disorders) | 2 (2) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-CsA treatment plus SoC (SAF) (N=32) | SoC alone (SAF) (N=30)
COVID-19 (Infections and infestations) | 7 (9) | 5 (5)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (7) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 2 (2)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Oedema peripheral (General disorders) | 3 (3) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-02-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT03657342/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-08): https://cdn.clinicaltrials.gov/large-docs/42/NCT03657342/SAP_001.pdf